CLINICAL TRIAL: NCT05547204
Title: Impact of Coffeeberry Extract on Skill Performance During Simulated Match Play in Academy Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2114
Record Dates: First submitted 2022-09-13; First posted 2022-09-21 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Skill Performance; Soccer Performance; Coffeeberry Effects
Keywords: coffeeberry; caffeine; polyphenols; chlorogenic acid; exercise; soccer; football; skill; performance
MeSH Terms: conditions — Motor Activity | interventions — Beverages

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coffeeberry beverage (Experimental): 300 ml drink containing 300 mg coffeeberry extract
  Interventions: Other: Beverage
- Color and flavor matched beverage (Placebo Comparator): 300 ml drink (0 mg coffeeberry extract, 0 mg caffeine)
  Interventions: Other: Beverage

INTERVENTIONS:
Other: Beverage — Free from added carbohydrates (contain 1g CHO only) and electrolytes are absent.

SUMMARY:
This study of soccer skill performance has three objectives:

1. Compare effects of coffeeberry (300mg) and placebo ingestion on dribbling speed and precision, passing speed and accuracy, and sprint speed during a full simulated soccer match.
2. Compare effects of coffeeberry (300mg) and placebo ingestion on subjective measures (mental / physical energy and activation-deactivation (feelings or mood) during a full simulated soccer match.
3. Compare effects of coffeeberry (300mg) and placebo ingestion on chlorogenic acid (CGA) and caffeine metabolites in the blood 1-hour post ingestion, and other blood metabolites (glucose/lactate) throughout the simulated soccer match.

ELIGIBILITY:
Inclusion Criteria:

* Provide valid informed consent prior to any study procedure
* Male soccer players age 16 to 28 years.
* >= 5-year soccer playing experience
* >= 1-year regularly soccer training
* Free of injuries
* Willing to avoid alcohol in the 48-h period prior to all visits
* Willing to avoid caffeinated products and apples, berries/cherries for 24-h prior to all visits
* Willing to record food intake over the 48-h period prior to the first trial and replicate for second trial
* Willing to abstain from strenuous physical activity for 24-h before all visits

Exclusion Criteria:

* Smoking
* Cardiovascular diseases
* Diabetes or other metabolic disease • Hypertension (>140/>90 mm Hg)
* Presence of injuries
* Major illnesses or surgery in prior 90 days
* Participation in another clinical trial in the past month

Ages: 16 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2022-12-04 (Actual)

PRIMARY OUTCOMES:
Dribbling speed | Change from pre-dose baseline through end of match 3.5 hours post consumption at multiple intervals each half of match
  m/sec, increase would be better. Simulated soccer match in an indoor gym with pre-set targets.
Dribbling precision | Change from pre-dose baseline through end of match 3.5 hours post consumption at multiple intervals each half of match
  Meters, more accuracy would be better. Simulated soccer match in an indoor gym with pre-set targets.
Passing accuracy | Change from pre-dose baseline through end of match 3.5 hours post consumption at multiple intervals each half of match.
  1 to 10 scale, a higher score would be better. Simulated soccer match in an indoor gym with pre-set targets.
Passing speed | Change from pre-dose baseline through end of match 3.5 hours post consumption at multiple intervals each half of match
  km/h, increased passing speed would be better. Simulated soccer match in an indoor gym with pre-set targets.
Sprint speed. | Change from pre-dose baseline through end of match 3.5 hours post consumption at multiple intervals each half of match
  m/sec, increased sprint speed would be better. In indoor gym with marked course.

SECONDARY OUTCOMES:
Blood analyte: Chlorogenic acid (CGA) | Pre-dose baseline, 60 minutes post-dose, half-time, and end of match (3.5 hours)
  mmol/L to evaluate primary outcomes. n.a. for placebo. Capillary blood draw for frozen plasma analysis
Blood analyte: Caffeine metabolites | Pre-dose baseline, 60 minutes post-dose, half-time, and end of match (3.5 hours)
  ug/ml, to evaluate primary outcomes. n.a. for placebo. Capillary blood draw for frozen plasma analysis
Blood analyte: Glucose | Pre-dose baseline, 60 minutes post-dose, half-time, and end of match (3.5 hours)
  mmol/L, more regulated would be better. Capillary blood draw for frozen plasma analysis
Blood analyte: Lactate | Pre-dose baseline, 60 minutes post-dose, half-time, and end of match (3.5 hours)
  mmol/L, lower (delayed rise) would be better. Capillary blood draw for frozen plasma analysis
Rating of perceived exertion (RPE) | Half-time and end of match (3.5 hours)
  By Borg scale, rated 6 to 20, very very light to very very hard. Lower values would be better
Activation-deactivation (feelings or mood) | Pre-dose baseline, 60 minutes post-dose, half-time, and end of match (3.5 hours)
  Checklist of 20 feelings using a 4 point scale from definitely do feel to definitely don't feel. More relaxed feelings or in a better mood would be better.
Mental energy | Pre-dose baseline, 60 minutes post-dose, half-time, and end of match (3.5 hours)
  Visual Analog Scale (VAS), vertical marking on 100 mm horizontal line. Higher energy would be better
Physical energy | Pre-dose baseline, 60 minutes post-dose, half-time, and end of match (3.5 hours)
  Visual Analog Scale (VAS), vertical marking on 100 mm horizontal line. Higher energy would be better
Gut comfort | Pre-dose baseline, 60 minutes post-dose, half-time, and end of match (3.5 hours)
  Visual Analog Scale (VAS), vertical marking on 100 mm horizontal line. No or less nausea, fullness or bloating would be better
Heart rate | Continuous from pre-dose baseline through end of match (3.5 hours)
  By electronic reading. Lower would be better.
Hydration status | Pre-dose baseline and end of match (3.5 hours)
  Urine osmolality in mOsm/kg change in concentration pre- vs. post-exercise

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Galloway, PhD, Principal Investigator — U. Stirling, Scotland
Locations (1):
- U. Stirling, Health Science and Sport, Stirling, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No